CLINICAL TRIAL: NCT02341859
Title: Lens Fitting Evaluation of CooperVision MyDay™ Compared With 1-DAY ACUVUE® TruEye® and DAILIES TOTAL1®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: JP-MKTG-201501
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- stenfilcon A and delefilcon A (Active Comparator): Participants randomized wear the stenfilcon A and the delefilcon A contralaterally.
  Interventions: Device: stenfilcon A; Device: delefilcon A
- stenfilcon A and narafilcon A (Active Comparator): Participants randomized wear the stenfilcon A and the narafilcon A contralaterally
  Interventions: Device: stenfilcon A; Device: narafilcon A

INTERVENTIONS:
Device: stenfilcon A — contact lens
  Other Names: MyDay
Device: delefilcon A — contact lens
  Other Names: 1-DAY ACUVUE
  Arms: stenfilcon A and delefilcon A
Device: narafilcon A — contact lens
  Other Names: DAILIES TOTAL1
  Arms: stenfilcon A and narafilcon A

SUMMARY:
Lens Fitting Evaluation of CooperVision MyDay™ Compared with 1-DAY ACUVUE® TruEye® and DAILIES TOTAL1®

DETAILED DESCRIPTION:
The aim of this non-dispensing study is to evaluate the fitting performance of MyDay™ 8.4 base curve, especially for flatter corneas, and compared it with 1-DAY ACUVUE® TruEye® 9.0 base curve and DAILIES TOTAL1® 8.8 base curve in a range of spherical powers.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft spherical contact lens wearer
* Has a contact lens spherical prescription between -4.00 to - 6.00 and higher than -7.00D (Diopters) (inclusive)
* Has a BFS (Best Fit Sphere) that is higher than 8.2 measured and calculated by corneal topography
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Patient contact lens refraction should fit within the available parameters of the study lenses
* Is willing to comply with the wear schedule
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Is not a habitual wearer of soft spherical contact lenses
* Has a contact lens prescription outside the range of the available parameters of the study lenses
* Has a contact lens prescription outside the range of the inclusion power range
* Has a spectacle cylinder ≥1.00D of cylinder in either eye
* Has a history of not achieving comfortable contact lens wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye
* Presence of clinically significant (grade > 2) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Moderate to severe dry eye
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses
* Has undergone corneal refractive surgery
* Is participating in any other type of eye related clinical or research study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD PhD, Principal Investigator — CRC-UC Berkeley
Locations (1):
- Clinical Research Center, University of California, Berkeley, Berkeley, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants enrolled in the study did not meet inclusion criteria. One participant was disqualified due to high power. All three participants therefore discontinued before lens randomization.
Groups:
- Stenfilcon A/Delefilcon A, Then Stenfilcon A/Narafilcon A: Participants randomized wear the stenfilcon A and delefilcon A lens pair contralaterally, and then cross over to wear the stenfilcon A and narafilcon A lens pair contralaterally.
  stenfilcon A: contact lens
  delefilcon A: contact lens
  narafilcon A: contact lens
- Stenfilcon A/Narafilcon A, Then Stenfilcon A/Delefilcon A: Participants randomized wear the stenfilcon A and narafilcon A lens pair contralaterally, and then cross over to wear the stenfilcon A and delefilcon A lens pair contralaterally.
  stenfilcon A: contact lens
  narafilcon A: contact lens
  delefilcon A: contact lens
Period: First Intervention (1 Day)
Arm/Group | Stenfilcon A/Delefilcon A, Then Stenfilcon A/Narafilcon A | Stenfilcon A/Narafilcon A, Then Stenfilcon A/Delefilcon A
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Stenfilcon A/Delefilcon A, Then Stenfilcon A/Narafilcon A | Stenfilcon A/Narafilcon A, Then Stenfilcon A/Delefilcon A
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participant Flow: Participants randomized wear the stenfilcon A and the delefilcon A contralaterally or the stenfilcon A and the narafilcon A contralaterally
  stenfilcon A: contact lens
  delefilcon A: contact lens
  narafilcon A: contact lens
Arm/Group | Overall Participant Flow
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (5.84)
Age, Continuous [Median (Full Range); unit: years] | 22 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Staining - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Conjunctival staining for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Scale 0-4, 0.5 steps 0=normal, 4=severe) N - nasal, T - temporal, S - superior, I - interior
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stenfilcon A (Delefilcon A Group); Delefilcon A: Participants randomized wear the stenfilcon A and the delefilcon A contralaterally.
  stenfilcon A: contact lens
  delefilcon A: contact lens
- Stenfilcon A (Narafilcon A Group): Participants randomized wear the stenfilcon A and the narafilcon A contralaterally
  stenfilcon A: contact lens
  narafilcon A: contact lens
- Narafilcon A: Participants randomized wear the stenfilcon A and the narafilcon A contralaterally.
  stenfilcon A: contact lens
  narafilcon A: contact lens
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  N | 0.42 (0.48) | 0.53 (0.51) | 0.68 (0.53) | 0.47 (0.49)
  T | 0.39 (0.43) | 0.34 (0.50) | 0.34 (0.37) | 0.45 (0.44)
  S | 0.13 (0.23) | 0.16 (0.24) | 0.21 (0.30) | 0.21 (0.30)
  I | 0.26 (0.26) | 0.18 (0.34) | 0.24 (0.35) | 0.34 (0.37)

2. Primary Outcome: Conjunctival Staining - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Conjunctival staining for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-4, 0.5 steps 0=normal, 4=severe) N - nasal, T - temporal, S - superior, I - interior
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Delefilcon A: Participants randomized wear the stenfilcon A and the delefilcon A contralaterally
  stenfilcon A: contact lens
  delefilcon A: contact lens
- Stenfilcon A (Narafilcon A Group); Narafilcon A: Participants randomized wear the stenfilcon A and the narafilcon A contralaterally.
  stenfilcon A: contact lens
  narafilcon A: contact lens
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  N | 0.97 (0.49) | 0.79 (0.54) | 1.00 (0.75) | 1.29 (0.87)
  T | 1.11 (0.74) | 0.47 (0.46) | 1.39 (0.89) | 0.97 (0.68)
  S | 0.26 (0.45) | 0.24 (0.31) | 0.45 (0.60) | 0.61 (1.04)
  I | 0.53 (0.56) | 0.63 (0.60) | 0.87 (0.60) | 1.24 (1.03)

3. Primary Outcome: Conjunctival Indentation - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Conjunctival indentation for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Scale 0-4, 0.5 steps 0=normal, 4=severe) N - nasal, T - temporal, S - superior, I - interior
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  N | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.08 (0.34)
  T | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  S | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  I | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.08 (0.34)

4. Primary Outcome: Conjunctival Indentation - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Conjunctival indentation for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-4, 0.5 steps 0=normal, 4=severe) N - nasal, T - temporal, S - superior, I - interior
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  N | 0.05 (0.16) | 0.16 (0.34) | 0.26 (0.45) | 0.08 (0.34)
  T | 0.18 (0.38) | 0.05 (0.16) | 0.53 (0.70) | 0.11 (0.36)
  S | 0.11 (0.32) | 0.00 (0.00) | 0.21 (0.45) | 0.21 (0.45)
  I | 0.16 (0.34) | 0.11 (0.27) | 0.21 (0.35) | 0.13 (0.33)

5. Primary Outcome: Limbal Redness - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Limbal redness for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Scale 0-4, 0.5 steps 0=normal, 4=severe)
  N - nasal, T - temporal, S - superior, I - interior
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  N | 0.97 (0.49) | 1.05 (0.44) | 0.97 (0.46) | 1.11 (0.70)
  T | 0.74 (0.35) | 0.89 (0.59) | 0.79 (0.67) | 0.97 (0.70)
  S | 0.82 (0.45) | 0.84 (0.50) | 0.79 (0.67) | 0.76 (0.63)
  I | 0.68 (0.45) | 0.63 (0.47) | 0.66 (0.41) | 0.71 (0.51)

6. Primary Outcome: Limbal Redness - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Limbal redness for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-4, 0.5 steps 0=normal, 4=severe) N - nasal, T - temporal, S - superior, I - interior
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  N | 1.08 (0.63) | 1.03 (0.35) | 1.05 (0.50) | 1.34 (0.76)
  T | 1.00 (0.44) | 1.03 (0.49) | 1.16 (0.55) | 1.13 (0.64)
  S | 0.89 (0.52) | 0.84 (0.44) | 0.84 (0.55) | 0.84 (0.50)
  I | 0.89 (0.49) | 0.84 (0.41) | 0.95 (0.64) | 0.95 (0.44)

7. Primary Outcome: Corneal Staining Type - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal staining type (ocular response) for for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Scale 0-4, 0.5 steps, 0=normal, 4=severe) C - central, N - nasal, T- temporal, S - superior, I - interior
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  C | 0.16 (0.47) | 0.05 (0.23) | 0.08 (0.34) | 0.00 (0.00)
  N | 0.34 (0.60) | 0.55 (0.86) | 0.53 (0.77) | 0.37 (0.70)
  T | 0.24 (0.45) | 0.34 (0.62) | 0.21 (0.45) | 0.32 (0.56)
  S | 0.45 (0.64) | 0.29 (0.51) | 0.45 (0.55) | 0.45 (0.50)
  I | 0.26 (0.48) | 0.37 (0.60) | 0.55 (0.76) | 0.53 (0.74)

8. Primary Outcome: Corneal Staining Type - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal staining type (ocular response) for for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-4, 0.5 steps, 0=normal, 4=severe) C - central, N - nasal, T- temporal, S - superior, I - interior
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  C | 0.00 (0.00) | 0.08 (0.34) | 0.00 (0.00) | 0.03 (0.11)
  N | 0.05 (0.23) | 0.08 (0.34) | 0.08 (0.34) | 0.71 (1.25)
  T | 0.18 (0.80) | 0.00 (0.00) | 0.21 (0.54) | 0.18 (0.61)
  S | 0.53 (0.59) | 0.74 (1.01) | 0.76 (0.84) | 0.47 (0.66)
  I | 0.26 (0.51) | 0.39 (0.86) | 0.71 (0.93) | 0.61 (0.68)

9. Primary Outcome: Corneal Staining Extent - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal staining extent (ocular response) for for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Scale 0-4, 0.5 steps, 0=normal, 4=severe) C - central, N - nasal, T- temporal, S - superior, I - interior
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  C | 0.13 (0.47) | 0.03 (0.11) | 0.03 (0.11) | 0.00 (0.00)
  N | 0.24 (0.51) | 0.34 (0.53) | 0.32 (0.53) | 0.24 (0.45)
  T | 0.13 (0.23) | 0.18 (0.42) | 0.18 (0.42) | 0.24 (0.42)
  S | 0.18 (0.25) | 0.16 (0.29) | 0.24 (0.31) | 0.32 (0.42)
  I | 0.24 (0.45) | 0.32 (0.71) | 0.37 (0.55) | 0.34 (0.47)

10. Primary Outcome: Corneal Staining Extent - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal staining extent (ocular response) for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-4, 0.5 steps, 0=normal, 4=severe) C - central, N - nasal, T- temporal, S - superior, I - interior
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  C | 0.00 (0.00) | 0.03 (0.11) | 0.00 (0.00) | 0.05 (0.23)
  N | 0.11 (0.46) | 0.03 (0.11) | 0.03 (0.11) | 0.24 (0.39)
  T | 0.03 (0.11) | 0.00 (0.00) | 0.09 (0.19) | 0.11 (0.32)
  S | 0.29 (0.30) | 0.29 (0.30) | 0.37 (0.37) | 0.29 (0.42)
  I | 0.18 (0.34) | 0.16 (0.29) | 0.37 (0.52) | 0.39 (0.43)

11. Primary Outcome: Corneal Staining Depth - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal staining depth for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group A assessed at baseline. (Scale 0-4, 0.5 steps, 0=normal, 4=severe) C - central, N - nasal, T- temporal, S - superior, I - interior
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  C | 0.11 (0.32) | 0.05 (0.23) | 0.05 (0.23) | 0.00 (0.00)
  N | 0.26 (0.45) | 0.34 (0.53) | 0.37 (0.50) | 0.26 (0.45)
  T | 0.26 (0.45) | 0.26 (0.45) | 0.21 (0.42) | 0.26 (0.45)
  S | 0.37 (0.50) | 0.26 (0.45) | 0.42 (0.51) | 0.47 (0.51)
  I | 0.26 (0.45) | 0.32 (0.48) | 0.42 (0.51) | 0.42 (0.51)

12. Primary Outcome: Corneal Staining Depth - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal staining depth (ocular response) for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-4, 0.5 steps, 0=normal, 4=severe) C - central, N - nasal, T- temporal, S - superior, I - interior
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  C | 0.00 (0.00) | 0.05 (0.23) | 0.00 (0.00) | 0.05 (0.23)
  N | 0.05 (0.23) | 0.05 (0.33) | 0.05 (0.23) | 0.32 (0.48)
  T | 0.05 (0.23) | 0.00 (0.00) | 0.16 (0.37) | 0.11 (0.32)
  S | 0.53 (0.51) | 0.55 (0.69) | 0.58 (0.51) | 0.42 (0.51)
  I | 0.26 (0.45) | 0.26 (0.45) | 0.47 (0.51) | 0.53 (0.51)

13. Primary Outcome: Corneal Shape Change - Tangential Radius - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal shape change for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at 6 hours by the topographer measurement and functions (map function of Tangential Curvature Map)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
mm | -0.007 (0.036) | -0.004 (0.080) | 0.009 (0.035) | 0.017 (0.027)

14. Primary Outcome: Corneal Shape Change - Wavefront Error - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Corneal shape change for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at 6 hours by the topographer measurement and functions (Wavefront Error Map)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
microns | 0.004 (0.022) | -0.006 (0.149) | -0.006 (0.024) | 0.004 (0.019)

15. Primary Outcome: Lens Fit - Corneal Coverage - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation for corneal coverage on insertion for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline with a 'yes' or 'no'.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Yes | 19 | 19 | 19 | 19
  No | 0 | 0 | 0 | 0

16. Primary Outcome: Lens Fit - Corneal Coverage - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation for corneal coverage on removal for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours with a 'yes' or 'no'.
Time Frame: 6 hours
Measure: Number; unit: participants
Groups:
- Stenfilcon A (Delefilcon A Group); Delefilcon A: Participants randomized wear the stenfilcon A and the delefilcon A contralaterally
  stenfilcon A: contact lens
  delefilcon A: contact lens
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Yes | 19 | 19 | 19 | 18
  No | 0 | 0 | 0 | 1

17. Primary Outcome: Lens Fit - Horizontal Centration - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of horizontal centration on insertion for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Temporal, Little temporal, Centered, Little nasal, Nasal)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Temporal | 0 | 0 | 0 | 2
  Little temporal | 2 | 0 | 0 | 4
  Centered | 17 | 19 | 19 | 13
  Little loose | 0 | 0 | 0 | 0
  Loose | 0 | 0 | 0 | 0

18. Primary Outcome: Lens Fit - Horizontal Centration - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of horizontal centration on removal for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Temporal, Little temporal, Centered, Little nasal, Nasal)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Temporal | 0 | 0 | 0 | 2
  Little temporal | 2 | 1 | 0 | 3
  Centered | 17 | 18 | 19 | 14
  Little loose | 0 | 0 | 0 | 0
  Loose | 0 | 0 | 0 | 0

19. Primary Outcome: Lens Fit - Vertical Centration - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of vertical centration on insertion for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Up, Little up, Centered, Little low, Low)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Up | 0 | 0 | 0 | 0
  Little Up | 0 | 0 | 0 | 1
  Centered | 15 | 16 | 17 | 10
  Little low | 3 | 3 | 2 | 6
  Low | 1 | 0 | 0 | 2

20. Primary Outcome: Lens Fit - Vertical Centration - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of vertical centration on removal for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Up, Little up, Centered, Little low, Low)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Up | 0 | 0 | 0 | 0
  Little Up | 0 | 0 | 0 | 0
  Centered | 18 | 18 | 18 | 10
  Little low | 0 | 1 | 1 | 3
  Low | 1 | 0 | 0 | 6

21. Primary Outcome: Lens Fit - Post-blink Movement - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of post-blink movement on insertion for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Tight, Little tight, Optimal, Little loose, Loose)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Tight | 0 | 0 | 0 | 0
  Little tight | 0 | 0 | 0 | 0
  Optimal | 18 | 18 | 18 | 19
  Little loose | 0 | 1 | 0 | 0
  Loose | 1 | 0 | 1 | 0

22. Primary Outcome: Lens Fit - Post-blink Movement - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of post-blink movement on removal for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Tight, Little tight, Optimal, Little loose, Loose)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Tight | 0 | 0 | 0 | 0
  Little tight | 0 | 0 | 0 | 0
  Optimal | 17 | 18 | 18 | 19
  Little loose | 2 | 1 | 1 | 0
  Loose | 0 | 0 | 0 | 0

23. Primary Outcome: Lens Fit - Tightness on up Gaze Blink Lag - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of tightness on up gaze blink lag for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline (insertion). (Optimal, Acceptable, No lag, Falls from cornea)
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Narafilcon A: Participants randomized wear the stenfilcon A and the narafilcon A contralaterally
  stenfilcon A: contact lens
  narafilcon A: contact lens
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Optimal | 12 | 14 | 16 | 11
  Acceptable | 6 | 5 | 3 | 5
  No lag | 0 | 0 | 0 | 0
  Falls from cornea | 1 | 0 | 0 | 3

24. Primary Outcome: Lens Fit - Tightness on up Gaze Blink Lag - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation of tightness on up gaze blink lag for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours on removal. (Optimal, Acceptable, No lag, Falls from cornea)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Optimal | 16 | 17 | 17 | 13
  Acceptable | 3 | 2 | 2 | 4
  No lag | 0 | 0 | 0 | 0
  Falls from cornea | 0 | 0 | 0 | 2

25. Primary Outcome: Lens Fit Overall - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation overall for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline. (Optimal, Almost optimal, Border line to wear, Not acceptable (cannot wear)).
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Optimal | 15 | 18 | 18 | 13
  Almost optimal | 4 | 1 | 1 | 5
  Border line to wear | 0 | 0 | 0 | 1
  Not acceptable (cannot wear) | 0 | 0 | 0 | 0

26. Primary Outcome: Lens Fit Overall - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Lens fit evaluation overall for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Optimal, Almost optimal, Border line to wear, Not acceptable (cannot wear)).
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  Optimal | 18 | 18 | 19 | 13
  Almost optimal | 1 | 1 | 0 | 4
  Border line to wear | 0 | 0 | 0 | 2
  Not acceptable (cannot wear) | 0 | 0 | 0 | 0

27. Secondary Outcome: Pain and Foreign Body Sensation (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of pain and foreign body sensation for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at baseline. 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  None | 18 | 16 | 12 | 9
  Mild | 1 | 3 | 5 | 8
  Moderate | 0 | 0 | 2 | 1
  Severe | 0 | 0 | 0 | 1

28. Secondary Outcome: Pain and Foreign Body Sensation (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of pain and foreign body sensation for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at 6 hours. 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  None | 15 | 15 | 13 | 11
  Mild | 2 | 3 | 6 | 7
  Moderate | 2 | 1 | 0 | 1
  Severe | 0 | 0 | 0 | 0

29. Secondary Outcome: Itching Sensation on Insertion (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of itching sensation on insertion for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at baseline. 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  None | 15 | 17 | 18 | 16
  Mild | 4 | 2 | 1 | 3
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

30. Secondary Outcome: Itching Sensation on Removal (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of itching sensation on removal for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at 6 hours. 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  None | 15 | 16 | 15 | 14
  Mild | 4 | 3 | 3 | 4
  Moderate | 0 | 0 | 1 | 1
  Severe | 0 | 0 | 0 | 0

31. Secondary Outcome: Red Eye (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of red eye on removal for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group is assessed at 6 hours. 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe)
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
participants
  None | 19 | 19 | 17 | 16
  Mild | 0 | 0 | 2 | 3
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

32. Secondary Outcome: Dryness (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of dryness for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline, 3 hours, and 6 hours. (Scale 0-100, 0=cannot wear, 100= no dryness).
Time Frame: Baseline, 3 hours, 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  Baseline | 91.3 (13.7) | 92.5 (14.2) | 93.0 (8.1) | 90.2 (11.5)
  3 hours | 87.8 (12.6) | 87.2 (16.0) | 89.7 (15.2) | 87.2 (19.0)
  6 hours | 88.7 (15.1) | 88.6 (14.9) | 85.4 (16.5) | 84.6 (120.3)

33. Secondary Outcome: Comfort (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of comfort for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline, 3 hours, and 6 hours. (Scale 0-100, 0=cannot wear, 100= no lens feeling).
Time Frame: Baseline, 3 hours, 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  Baseline | 90.0 (11.8) | 92.7 (8.2) | 84.3 (20.6) | 84.6 (14.4)
  3 hours | 90.0 (16.3) | 88.4 (17.2) | 90.2 (12.5) | 86.1 (17.7)
  6 hours | 86.1 (16.8) | 88.4 (14.4) | 88.1 (13.9) | 85.6 (17.8)

34. Secondary Outcome: Handling (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of handling for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline (ease of insertion) and 6 hours (ease of removal). (Scale 0-100, 0=cannot handle at all, 100=no problem at all).
Time Frame: Baseline and 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  Baseline (insertion) | 95.8 (5.3) | 93.0 (9.4) | 90.9 (10.8) | 91.3 (12.8)
  6 hours (removal) | 81.6 (27.7) | 86.4 (22.5) | 88.3 (21.0) | 93.2 (19.1)

35. Secondary Outcome: Vision (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of vision for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at baseline, 3 hours, and 6 hours. (Scale 0-100, 0=cannot see due to blur vision, 100=clear vision without any blur image).
Time Frame: Baseline, 3 hours, 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale
  Baseline | 90.0 (13.6) | 94.1 (6.9) | 86.5 (19.1) | 90.6 (7.7)
  3 hours | 93.5 (11.4) | 96.8 (3.9) | 93.2 (10.0) | 90.3 (13.0)
  6 hours | 93.0 (8.1) | 93.9 (9.5) | 92.4 (7.0) | 90.5 (9.7)

36. Secondary Outcome: Overall Wearing Satisfaction (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of overall wearing satisfaction for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Scale 0-100, 0=very poor, 100=very satisfied).
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale | 86.5 (17.4) | 88.6 (14.4) | 86.8 (13.4) | 83.4 (17.5)

37. Secondary Outcome: Lens Preferences (Subjective Rating) - Stenfilcon A/Delefilcon A and Stenfilcon A/Narafilcon A
Description: Subjective ratings of lens preferences for stenfilcon A/delefilcon A group and stenfilcon A/narafilcon A group assessed at 6 hours. (Which lens is preferred)
Time Frame: 6 hours
Population: Preference is missing for 1 participant in the stenfilcon A/delefilcon A group whom did not answer preference question of which lens is preferred.
Measure: Number; unit: participants
Arm/Group | Stenfilcon A (Delefilcon A Group) | Delefilcon A | Stenfilcon A (Narafilcon A Group) | Narafilcon A
Number analyzed (Participants) | 18 | 18 | 19 | 19
participants | 7 | 11 | 15 | 4

ADVERSE EVENTS:
Groups:
- Stenfilcon A: Participants randomized wear the stenfilcon A and the delefilcon A contralaterally or the stenfilcon A and the narafilcon A contralaterally
  stenfilcon A: contact lens
  delefilcon A: contact lens
  narafilcon A: contact lens
Arm/Group | Stenfilcon A | Delefilcon A | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.